CLINICAL TRIAL: NCT06396234
Title: Pilot Study Comparing Intubation Via Video Laryngeal Mask Airways (VLMAs) Versus Video Laryngoscopy: Efficacy and Patient Outcomes in General Anesthesia Procedures
Brief Title: Study Comparing Intubation Via Video Laryngeal Mask Airways (VLMAs) Versus Video Laryngoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never approved by the IRB. Was not initiated
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-15294
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Laryngeal Mask Airways; Airway Management; Supraglottic Airways; Video-assisted
MeSH Terms: interventions — Airway Management

STUDY DESIGN:
Intervention Model Description: Single-centered, Randomized, Pilot Study
Who Masked: Participant
Masking Description: Participant will have agreed to the study and randomized device or technique will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Safe VLM (Experimental): The device will be placed after patient is anesthetized. Following placement, the glottis will be observed and endotracheal tube will be placed.
  Interventions: Device: Safe VLM and airway management
- Video laryngoscopy (Active Comparator): Following anesthetic induction, endotracheal intubation will be performed with a video laryngoscope.
  Interventions: Procedure: Endotracheal intubation using video laryngoscope
- SaCo VLM (Experimental): The device will be placed after patient is anesthetized. Following placement, the glottis will be observed and endotracheal tube will be placed.
  Interventions: Device: SaCo VLM and airway management

INTERVENTIONS:
Device: Safe VLM and airway management — Once the device is placed, following assessment, endotracheal intubation will be performed via the device.
  Other Names: SafeLM® Video Laryngeal Mask System by Magill Medical Technology Co. Ltd
  Arms: Safe VLM
Procedure: Endotracheal intubation using video laryngoscope — Endotracheal intubation (size 7.0 mm) using video laryngoscope
  Arms: Video laryngoscopy
Device: SaCo VLM and airway management — Once the device is placed, following assessment, endotracheal intubation will be performed via the device.
  Other Names: SaCo (UESCOPE® 2) by UE Medical Devices, Inc.
  Arms: SaCo VLM

SUMMARY:
The goal of this clinical trial is to compare the overall performance and patient outcomes of two video-assisted laryngeal mask airways (VLMAs) devices called Safe and Comfortable (SaCo) VLM and SafeLM® (Safe VLM) versus video laryngoscopy for airway management in adult patients, without an anticipated difficult airway, that are undergoing elective general anesthesia procedures.

The main question it aims to answer is: Can both VLMAs improve patient-centered outcomes in the perioperative and postoperative periods in comparison to endotracheal tube (ETT) intubation? Thirty participants will undergo randomized VLMA with either the Safe VLM (15 participants) or the SaCo VLM (15 participants). And 15 participants will be intubated with ETT using video laryngoscopy, as the control group. Researchers will evaluate the efficacy of these two video-assisted devices in adult patients without an anticipated difficult airway in elective general anesthesia procedures. Other patient outcomes and exploratory endpoints will be recorded as well.

DETAILED DESCRIPTION:
INVESTIGATIONAL DEVICES NAMES SaCo® (UESCOPE® 2) by UE Medical Devices, Inc SafeLM® Video Laryngeal Mask System by Magill Medical Technology Co. Ltd

STUDY RATIONALE New airway devices for anesthesiology are constantly being developed to improve patient overall safety, reduce perioperative risks and complications, enhance recovery, and prevent postoperative adverse-related outcomes. The first and second generation supraglottic airway devices (SADs) have satisfactory features which provide an effective airway and ventilation without the need for more aggressive endotracheal intubation. Nevertheless, these are inserted in a "blind" fashion; malpositioning and potential airway compromise occurs in 50-80% of placements.

Thus, direct vision-guided placement using newer third generation video laryngeal mask airways (VLMAs), can ensure optimal positioning, adequate lung ventilation, and perioperative real-time visualization of the airway. This allows for assessment and any needed corrective maneuvers if they become necessary. The two types of FDA-approved VLMAs that this study will test are: 1) the SafeLM® Video Laryngeal Mask System, which has a camera angle-adjusting handle that allows direct vision up to 140° angle of view of the oropharynx and larynx, with a monitor that is embedded in the device; and 2) the SaCo® Video Laryngeal Mask, which has an embedded camera fixed into the shaft of the device, which attaches to an external monitor. Both devices can guide endotracheal intubation through the ventilation channel under direct vision.

Recent studies have demonstrated the various applications of SaCo VLM for the management of difficult airways in adult patients requiring general anesthesia. This pilot study will be a single-center randomized controlled trial of 45 healthy adult patients undergoing general anesthesia. We aim to explore the efficacy of both VLMAs and evaluate patient perioperative and postoperative outcomes; both are expected to replicate and, possibly, even improve on the outcomes from the conventional video laryngoscopy.

INVESTIGATIONAL DEVICE INTENDED USE The intended use of the video-guided LMAs is to aid in optimal placement of supraglottic airway devices, which will require additional ETT intubation, in participants without anticipated difficult airways.

NUMBER OF SITES One study site: Montefiore Medical Center

SUBJECT POPULATION The two devices will be studied in adult patients, without an anticipated difficult airway, presenting for elective general anesthesia and airway management.

NUMBER OF PARTICIPANTS Thirty participants will undergo supraglottic placement with either the SafeLM (15 participants) or the SaCo VLMAs (15 participants). Fifteen participants will be intubated with ETT via video laryngoscopy, as the control group.

STUDY OBJECTIVE To evaluate the efficacy of the two video-assisted supraglottic devices in elective adult patients without an anticipated difficult airway; other patient outcomes and exploratory endpoints will be recorded as well.

ELIGIBILITY:
Inclusion Criteria:

* Any sex
* Age ≥ 18 yrs
* BMI ≥ 40 kg/m2
* American Society of Anesthesiologists (ASA) class I-III
* With intention to undergo endotracheal intubation
* Understanding the purpose of the study and signing the informed consent

Exclusion Criteria:

* ASA IV
* History of upper respiratory infection within 2 weeks
* Presence of risk factors for gastric reflux or aspiration
* Symptomatic bronchial asthma
* Restricted mouth opening (﹤2 cm)
* Upper airway tumors, abscesses, foreign bodies or airway stenosis
* Requiring one-lung ventilation for thoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Successful first-attempt placement rate of VLMA | Intraoperative period, from the beginning of the general anesthesia induction to VLMA placement, up to 30 seconds
  The first-attempt success rate of VLMA device placement will be determined. Insertion will be considered successful if the VLMA is placed without any resistance and is confirmed to be optimally positioned based on the laryngeal mask visual screen, end-tidal carbon dioxide (CO2) after placement and ventilatory parameters. This will be reported as a dichotomous variable (successful vs unsuccessful).
Successful first-attempt placement rate of endotracheal intubation via video laryngoscopy | Intraoperative period, from the beginning of the general anesthesia induction to ETT placement, up to 45 seconds
  Insertion will be considered successful if the endotracheal tube slides through the VLMA without any resistance and is confirmed to be optimally positioned based on observation via the laryngeal mask visual monitor screen and capnography. This will be reported as a dichotomous variable (successful vs unsuccessful).
Number of participants with change in mean blood pressure by 20% from baseline mean blood pressure | Perioperative period, from the beginning of the general anesthesia induction to the end of evaluation, up to 1 day
  Measurement of blood pressure will be taken before and after intubation.
Number of participants with change in heart rate by 20% from baseline heart rate | Perioperative period, from the beginning of the general anesthesia induction to the end of evaluation, up to 1 day
  Measurement of heart rate will be taken before and after intubation.
Number of participants change in oxygen saturation by 20% from baseline | Perioperative period, from the beginning of the general anesthesia induction to the end of evaluation, up to 1 day
  Measurement of oxygen saturation will be taken before and after intubation.
Incidence of pharyngalgia, bleeding, hoarseness, and dysphagia events | Postoperative period at 1 hour and 24 hours after procedure
  Incidence of pharyngalgia, bleeding, hoarseness, and dysphagia events will be summarized as observed as reported by patients

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) | Postoperative period, up to one day following procedure
  Incidence of PONV events will be summarized as observed as reported by patients
Number of participants with postoperative hypertension by >30% of baseline, requiring treatment | Postoperative period, up to 1 hour
  Measurement of mean blood pressure will be taken and compared with baseline. If greater than 30%, participants will be given antihypertensive medication. The number/percentage of participants will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Irene Osborn, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gomez-Rios MA, Lopez T, Sastre JA, Gaszynski T, Van Zundert AAJ. Video laryngeal masks in airway management. Expert Rev Med Devices. 2022 Nov;19(11):847-858. doi: 10.1080/17434440.2022.2142558. Epub 2022 Nov 8. PMID 36308748
- [Result] Gordon J, Cooper RM, Parotto M. Supraglottic airway devices: indications, contraindications and management. Minerva Anestesiol. 2018 Mar;84(3):389-397. doi: 10.23736/S0375-9393.17.12112-7. Epub 2017 Oct 12. PMID 29027772
- [Result] Hussain D, Kundal R, Kumar A, Sabharwal N. An Analysis of the Comparative Efficacy Between a Third-Generation and a Second-Generation Supraglottic Airway Device in Patients Undergoing Laparoscopic Cholecystectomy. Cureus. 2022 Feb 25;14(2):e22592. doi: 10.7759/cureus.22592. eCollection 2022 Feb. PMID 35355545
- [Result] Lai CJ, Yeh YC, Tu YK, Cheng YJ, Liu CM, Fan SZ. Comparison of the efficacy of supraglottic airway devices in low-risk adult patients: a network meta-analysis and systematic review. Sci Rep. 2021 Jul 23;11(1):15074. doi: 10.1038/s41598-021-94114-7. PMID 34301986
- [Result] Sun Y, Huang L, Xu L, Zhang M, Guo Y, Wang Y. The Application of a SaCoVLMTM Visual Intubation Laryngeal Mask for the Management of Difficult Airways in Morbidly Obese Patients: Case Report. Front Med (Lausanne). 2021 Nov 18;8:763103. doi: 10.3389/fmed.2021.763103. eCollection 2021. PMID 34869469
- [Result] Timmermann A, Bergner UA, Russo SG. Laryngeal mask airway indications: new frontiers for second-generation supraglottic airways. Curr Opin Anaesthesiol. 2015 Dec;28(6):717-26. doi: 10.1097/ACO.0000000000000262. PMID 26539790
- [Result] Van Zundert AAJ, Gatt SP, Van Zundert TCRV, Kumar CM, Pandit JJ. Features of new vision-incorporated third-generation video laryngeal mask airways. J Clin Monit Comput. 2022 Aug;36(4):921-928. doi: 10.1007/s10877-021-00780-3. Epub 2021 Dec 17. PMID 34919170
- [Result] Van Zundert AAJ, Kumar CM, Van Zundert TCRV, Gatt SP, Pandit JJ. The case for a 3rd generation supraglottic airway device facilitating direct vision placement. J Clin Monit Comput. 2021 Apr;35(2):217-224. doi: 10.1007/s10877-020-00537-4. Epub 2020 Jun 15. PMID 32537697
- [Result] van Zundert AAJ, Wyssusek KH, Pelecanos A, Roets M, Kumar CM. A prospective randomized comparison of airway seal using the novel vision-guided insertion of LMA-Supreme(R) and LMA-Protector(R). J Clin Monit Comput. 2020 Apr;34(2):285-294. doi: 10.1007/s10877-019-00301-3. Epub 2019 Apr 5. PMID 30953222
- [Result] Van Zundert AA, Kumar CM, Van Zundert TC. Malpositioning of supraglottic airway devices: preventive and corrective strategies. Br J Anaesth. 2016 May;116(5):579-82. doi: 10.1093/bja/aew104. No abstract available. PMID 27106958
- [Result] Yan CL, Zhang YQ, Chen Y, Qv ZY, Zuo MZ. Comparison of SaCoVLM video laryngeal mask-guided intubation and i-gel combined with flexible bronchoscopy-guided intubation in airway management during general anesthesia: a non-inferiority study. BMC Anesthesiol. 2022 Sep 22;22(1):302. doi: 10.1186/s12871-022-01843-x. PMID 36138363
- [Result] Yan CL, Chen Y, Sun P, Qv ZY, Zuo MZ. Preliminary evaluation of SaCoVLM video laryngeal mask airway in airway management for general anesthesia. BMC Anesthesiol. 2022 Jan 3;22(1):3. doi: 10.1186/s12871-021-01541-0. PMID 34979936
- [Result] Zhi J, Deng XM, Zhang YM, Wei LX, Wang QY, Yang D. Preliminary evaluation of SaCoVLM video laryngeal mask-guided intubation in airway management for anesthetized children. BMC Anesthesiol. 2023 Feb 8;23(1):49. doi: 10.1186/s12871-023-01996-3. PMID 36755214